CLINICAL TRIAL: NCT04761796
Title: Prevalence and Factors Associated With Insomnia and Sleep Time in a Sample of Professional Flight Members
Brief Title: Sleep Time and Insomnia Factors Among Professional Flight Members
Acronym: SOMNAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A02069-30; NCT04761809 (obsolete NCT alias)
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Insomnia; Sleepiness
Keywords: Sleeping time; Chronic insomnia; Sleepiness; Flight members
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleepiness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Professional flight members
  Interventions: Other: Sleeping condition self-questionnaire

INTERVENTIONS:
Other: Sleeping condition self-questionnaire — Professional flight members will answer a self questionnaire related to their sleeping conditions

SUMMARY:
Sleep is a physiological function that plays an essential role in many somatic, cognitive or psychological processes. Although the criteria for sleep effectiveness are multiple, its quantity is unanimously recognized as a major determinant of health. Too little sleep time is indeed associated with an increase in metabolic, cardiovascular and accidental morbidity and mortality, caused by sleepiness during journeys or at the workplace. In the wake of recent work in the general French population, a specific study on the prevalence and factors associated with sleeping time and chronic insomnia among flight members appears relevant. Chronic insomnia and sleep debt can thus be assumed to be more common among aircrews than in the general population, due to these specific operational constraints. Better consideration of certain sleep disorders in professional flight members could make it possible to adapt prevention or countermeasures strategies intended to optimize risk management with regard to flight safety.

DETAILED DESCRIPTION:
Today, time dedicated to sleep is in competition with working time, transport time or time spent on new technologies, in a professional or recreational setting. Faced with the public health issue thus raised, studies have highlighted the interest of studying the relationships between sleep time and socio-demographic factors, beyond the mere implication of sleep pathologies. However, among these pathologies, the place of insomnia is not negligible: it is indeed the most frequent sleep disorder (16% of French people in 2010) and represents an important source of involuntary reduction in sleep time, likely to increase inappropriate sleepiness during periods of wakefulness, in the context of activities sometimes involving safety.

Flight crews are exposed to specific operational constraints, both in civilian and military environments, likely to compromise the recovery function of sleep (operational fatigue, extended working ranges, repetitions of time differences, etc.). These constraints, conducive to compromising the levels of vigilance and cognitive performance required, are also at risk of cardio-metabolic complications. They therefore raise the issue of controlling risks and maintaining aviation safety.

The issue of pilot fatigue remains an essential issue for the safety of flight operations. In the context of air transport, several determinants of operational fatigue have been identified, such as irregular sleep schedules, large, irregular and sometimes unpredictable activity ranges, sleep debts, night flights and circadian disturbances in connection with multiple and repeated changes of time zones. If these factors must deal within airlines with rules more often based on alternating "work / rest" than "sleep / wakefulness", the laws and regulations in force, within the aeronautical industry, are now oriented towards scientific approaches to the management of fatigue in commercial aviation, by emphasizing the importance of sleep and taking into account circadian rhythms.

Currently, the vast majority of studies devoted to the sleep of aviation flight personnel are therefore limited to the cases of commercial aviation airline pilots. They have established that most flights, especially over long-haul sectors, involve disturbances of the circadian rhythm, fractionation and restriction of sleep that are harmful to cognitive performance and the risk of accidents. Most publications have looked for associations between sleep measures and performance in an operational context. Some have been able to demonstrate that the classic methods of evaluating sleep in flight (by actimetric readings, sleep diaries or subjective evaluation of self-questionnaires) were correlated with reference data obtained by polysomnography, strongly for the duration of sleep but moderately to weakly for its effectiveness. In the specific case of sleep duration, self-report questionnaires have proven to be a reliable alternative to in-flight actimetric measurements.

The majority of studies have been designed considering pilot sleep as a determinant of in-flight performance, especially during long (12 to 16 hours) and very long (over 16 hours) flights. On the other hand, taking into account the consequences of aeronautical activity on the sleep of pilots is relatively rare in the scientific literature. Thus, most "ecological" studies, known as field studies, generally focus on specific flights with limited time slots and small sample sizes, limiting the scope of the results regarding the effects of flights on sleep. Currently, the main topic of interest is still the sleep of pilots immediately before, during and after duty periods, but without characterizing their baseline sleep, observed during periods of rest.

From this perspective, a study looked at the basic sleep of airline pilots, making comparisons to samples of the general North American population. On a total number of 332 long-haul pilots, the actimetric data revealed longer sleep times during rest periods, highlighting the influence of environmental stresses deemed to be risky to health. In addition, the influence of socio-demographic and professional parameters was reported in a study of 435 pilots. The high prevalence of sleep disorders, drowsiness and fatigue have been documented, as well as an increased risk of fatigue for flight crews on short and medium-haul flights, in connection with the working hours and repetition of rotations.

This study project therefore fits into this global context, in the light of 3 innovative perspectives:

* Target a rich and varied professional panel of aeronautical specialties (not limited to airline pilots only), integrating civil and military status, engaged in distinct operational frameworks but where risk control and aviation safety prevail;
* Recruit a large sample, without current equivalent to our knowledge in the scientific literature;
* Benefit from equivalent and recent data from a study carried out on a very large representative sample of the general French population

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 60 years of age
* Professional flight members
* All aeronautical specialties
* Going for an expert aeromedical visit
* Not opposing the study

Exclusion Criteria:

* Presenting himself/herself for a first medical exam
* Opposition to the study
* Under 18 years of age
* Non-professional aircrew
* Pregnant woman, parturient, breastfeeding
* Person deprived of liberty by a judicial or administrative decision, person undergoing psychiatric treatment by virtue of Articles L. 3212-1 and L. 3213-1 which do not fall under the provisions of Article L. 1121-8
* Adult person subject to a legal protection measure
* Person unable to express consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is composed of military aircrew.
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
To describe the average sleep time within a sample of the French professional flight members | 30 minutes
  Average total nighttime sleep time estimated using a self-administered questionnaire

SECONDARY OUTCOMES:
Chronic insomnia | 30 minutes
  Criteria of the International Classification of Sleep Disease (ICSD-3) of the American Academy of Sleep Medicine (items A, B and C of the questionnaire)
Subjective excessive sleepiness Subjective excessive sleepiness | 30 minutes
  Subjective excessive sleepiness will be estimated on the basis of the replies to the questionnaire : items of Epworth Sleepiness Scale (ESS). The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
Sleep duration, sleep debt, sleep restriction | 30 minutes
  Sleep duration, sleep debt, sleep restriction will be estimated on the basis of the replies to the questionnaire
Ideal sleep time | 30 minutes
  Ideal sleep time will be estimated on the basis of the replies to the questionnaire
Sociodemographic factors | 30 minutes
  Sociodemographic factors will be estimated on the basis of the replies to the questionnaire Predictive factors of sleep duration, sleepiness and chronic insomnia will be assessed using a top-down liner and/or logistic models taking into account socio-demographic variables
Aeronautical factors | 30 minutes
  Aeronautical factors will be estimated on the basis of the replies to the questionnaire Predictive factors of sleep duration, sleepiness and chronic insomnia will be assessed using a top-down liner and/or logistic models taking into account occupational variables

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Huiban, MD, Study Director — French Army Health Services
Locations (1):
- Cempn, Hia Sainte Anne, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No